CLINICAL TRIAL: NCT03975894
Title: A Feasibility Trial of Serial Prophylactic Exchange Blood Transfusion in Pregnant Women With Sickle Cell Disease Aiming to Improve Maternal and Infant Outcomes
Brief Title: TAPS2 Transfusion Antenatally in Pregnant Women With SCD
Acronym: TAPS2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other); Barts & The London NHS Trust (Other); The Whittington Hospital NHS Trust (Other Government); St Mary's NHS Trust (Other Government); University College London Hospitals (Other); St George's University Hospitals NHS Foundation Trust (Other); London School of Hygiene and Tropical Medicine (Other); King's College London (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAPS2version3
Record Dates: First submitted 2019-05-17; First posted 2019-06-05 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Sickle Cell Disease; Pregnancy, High Risk; Blood Transfusion Complication
Keywords: pregnancy; exchange transfusion; perinatal complications
MeSH Terms: conditions — Anemia, Sickle Cell; Transfusion Reaction

STUDY DESIGN:
Intervention Model Description: Regular prophylactic blood transfusion given every 6-10 weeks during pregnancy to maintain a HbS% of <30%
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Regular prophylactic blood transfusion given every 6-10 weeks during pregnancy to maintain a HbS% of <30%.
  Interventions: Biological: Serial prophylactic exchange blood transfusion (SPEBT).
- Control (No Intervention): Symptom directed blood transfusion during pregnancy.

INTERVENTIONS:
Biological: Serial prophylactic exchange blood transfusion (SPEBT). — Serial prophylactic exchange blood transfusion (SPEBT) will be given via automated apheresis technology. SPEBT will be carried out on the haematology day unit or on the antenatal day unit/ward in accordance with local policies in participating units. The procedure will be carried out using standard operating procedures, by the clinical or research nurse/midwife, haematology day unit staff or specialist sickle nursing staff. Venous access will be via peripheral access if possible or by femoral line access if not.
  SPEBT will be commenced between 6 and 18+0 weeks gestation. It will be repeated at 6-10 weekly intervals aiming to maintain HbS% <30%. It will continue throughout pregnancy and be stopped at the end of pregnancy.
  Number of red cell units used per transfusion will depend on patient weight and pre-transfusion HbS%, but will usually be between 6 and 8 units of red cells on each occasion of exchange transfusion.
  Arms: Intervention

SUMMARY:
Sickle Cell Disease (SCD) is a serious inherited blood disorder affecting red blood cells. When oxygen levels drop the red cells become abnormally shaped and unable to move through the blood vessels easily. Blood and oxygen do not reach body organs, resulting in episodes of severe pain and other complications. Pregnant women with SCD have an increased risk of both sickle and pregnancy complications, including raised blood pressure. Their babies may grow more slowly in the womb, are more likely to be born early and need special care, and have a higher risk of dying. The only treatments currently available for women with SCD are Hydroxycarbamide (which cannot be used during pregnancy) and blood transfusion. Currently, blood transfusion is only used during pregnancy to treat emergency complications. It has been suggested that giving blood transfusions throughout pregnancy could improve outcomes for both mother and babies. In Serial Prophylactic Exchange Blood Transfusion (SPEBT), sickle blood is mechanically removed and simultaneously replaced with donor red cells. A trial is needed to assess SPEBT given every 6-10 weeks, starting before 18 weeks of pregnancy, compared to standard care. This trial will evaluate outcomes for women (e.g. hospital admission, frequency of crisis) and their infants (e.g. early delivery, birthweight). However, the feasibility of such a study needs to be assessed before embarking on a large multicentre trial. This study is therefore a feasibility study in which we will randomly allocate participants to have either SPEBT or standard care. The study will be carried out in multiple maternity units in England and last two years. The willingness of eligible women to join the study will be assessed, along with how many participants remain part of the study until the end and if participants find the intervention acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with sickle cell disease (all genotypes)
* Gestation 18+0 weeks or below
* Willing and able to give informed consent
* Singleton pregnancy

Exclusion Criteria:

* On long term transfusion programme prior to pregnancy for amelioration of SCD
* Prior Hyperhaemolysis
* Red cell phenotype or antibodies present prevent likely provision of adequate red cell units to support elective EBT programme
* Unable to receive blood transfusion for social, religious or clinical reasons
* Current diagnosis of major medical or psychiatric comorbidity which in the randomising clinicians opinion renders them unable to enter trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  ratio of women eligible:women randomised

SECONDARY OUTCOMES:
Feasibility endpoints | up to 6 weeks postpartum
  Number of women eligible, reasons for refusal, rate and reasons for attrition, protocol adherence
Maternal hospital admissions | Every 6-8 weeks from enrolment to 6 weeks postpartum
  Antenatal and postnatal inpatient stays
Frequency and severity of painful crisis | Every 6-8 weeks from enrolment to 6 weeks postpartum
  self-reported symptoms (mild/moderate/severe/extremely severe) and use of opioid analgesics
Mode of birth | 40 weeks
SCD-related complications | Every 6-8 weeks from enrolment to 6 weeks postpartum
  E.g. acute chest syndrome, stroke, pre-eclampsia, venous thromboembolism.
Fetal demise/stillbirth | 40 weeks
Infant birthweight | 40 weeks
  Birthweight in grams
Gestation at birth | 40 weeks
  Gestation at birth in completed weeks and days
Fetal condition at birth | 40 weeks
  Apgar score at five minutes
Neonatal intensive care unit/critical care admission | 6 weeks postpartum
Safety outcome 1: transfusion reaction | Every 6-8 weeks from enrolment to 6 weeks postpartum
Safety outcome 2: Alloimmunisation | Every 6-8 weeks from enrolment to 6 weeks postpartum
  Irregular presence of red cell antibodies will be measured by routine blood test
Safety outcome 3: Delayed haemolytic transfusion reaction | Every 6-8 weeks from enrolment to 6 weeks postpartum
  After 7 days following transfusion:
  A. Fatigued, fever, jaundice, dark brown coca-cola urine B. Raised pulse, anaemia C. Dropping Haemoglobin, break down of haemoglobin, increased bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Oteng-Ntim, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Whittington Health NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oteng-Ntim E, Oakley LL, Robinson V, Brien S, Joseph J, Sharif J, McCabe L, Thompson H, Awogbade M, Johns J, Brunetta DM, Seed PT. Prophylactic exchange transfusion in sickle cell disease pregnancy: a TAPS2 feasibility randomized controlled trial. Blood Adv. 2024 Aug 27;8(16):4359-4369. doi: 10.1182/bloodadvances.2024012923. PMID 38954844
- [Derived] Oakley LL, Awogbade M, Brien S, Briley A, Chorozoglou M, Drasar E, Johns J, Rhodes E, Robinson V, Seed P, Sharif J, Singh C, Telfer P, Thompson H, Watt-Coote I, Howard J, Oteng-Ntim E. Serial prophylactic exchange blood transfusion in pregnant women with sickle cell disease (TAPS-2): study protocol for a randomised controlled feasibility trial. Trials. 2020 Apr 20;21(1):347. doi: 10.1186/s13063-020-4212-8. PMID 32312326